CLINICAL TRIAL: NCT02360644
Title: Drug Metabolizing Enzyme and Transporter Function in Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Pittsburgh (Other); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-1150; UL1TR001082 (NIH); 1R01GM107122-01A1 (NIH)
Record Dates: First submitted 2014-12-19; First posted 2015-02-10 (Estimated); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Chronic Kidney Diseases; Deficiency, Vitamin D
MeSH Terms: conditions — Renal Insufficiency, Chronic; Vitamin D Deficiency | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Drug Metabolism and Transport (Experimental): The aim of Arm 1 is to determine the effect of vitamin D deficiency and repletion on xenobiotic clearance in vivo. The study will evaluate the in vivo function of targeted metabolism and transport pathways in 40 CKD and 18 healthy volunteer subjects (controls) under the influence of a vitamin D depleted state and repeated under a vitamin D replete state with cholecalciferol.
  The function of two major phase I drug metabolizing enzymes (CYP2B6, CYP3A), and three transporters [P-gp, MRP2, and MATE1/2K] will be assessed by administering oral bupropion, midazolam, olmesartan, and fexofenadine.
  Interventions: Dietary Supplement: Cholecalciferol
- Arm 2: Vitamin D Pharmacokinetics (Experimental): The aim of Arm 2 is to determine the effect of CKD on the in vivo function of individual CYP450s responsible for vitamin D metabolism and their functional relevance on the pharmacokinetics of cholecalciferol. A total of 90 CKD subjects will be enrolled [30 per group: group I (CKD stage 1/2), group II (CKD stage 3), and group III (CKD stage 4/5, pre-ESRD)], as well as 30 healthy controls.
  Interventions: Dietary Supplement: Cholecalciferol

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — Vitamin D deficient patients, in both Arms, will be administered Cholecalciferol 5,000 IU daily.
  Other Names: Vitamin D

SUMMARY:
This study investigates the effect of vitamin D deficiency on drug metabolism and transport in patients with chronic kidney disease (CKD) and in healthy controls.

The central hypothesis is that vitamin D concentrations independently affect metabolism and transport function in CKD patients. An over-arching goal of this proposal is to make drug therapies safer and more effective to reduce the significant morbidity and mortality in patients with CKD.

DETAILED DESCRIPTION:
Specific Aim 1: Determine the effect of vitamin D deficiency and repletion on xenobiotic clearance in vivo. The study will mechanistically evaluate the function of major pathways of metabolism and transport by prospectively studying clearance phenotypes utilizing "probe" drugs commonly used for this purpose in CKD patients and healthy volunteers under vitamin D deficient and replete states. Bupropion, midazolam, olmesartan, fexofenadine, in addition to an endogenous probe (N-methylnicotinamide), will be used to phenotype major phase I drug metabolizing enzymes [cytochrome P450 2B6 (CYP2B6), cytochrome P450 3A4/5 (CYP3A4/5)], and transporters [multidrug resistance associated protein 2 (MRP2), P-glycoprotein (P-gp), and multidrug and toxin extrusion protein 1/2K (MATE1/2K)], respectively. Hypothesis: The in vivo function of individual pathways of xenobiotic metabolism and transport are affected by vitamin D status (and CKD).

Specific Aim 2: Determine the effect of CKD on the in vivo function of individual CYPs responsible for vitamin D metabolism and the pharmacokinetics of cholecalciferol (vitamin D3). The research will prospectively measure the activity of CYP450s responsible for cholecalciferol metabolism, and simultaneously evaluate the pharmacokinetics (PK) of cholecalciferol after single- and multiple-dose administration to CKD patients (stages 1-5) and healthy volunteers. Hypothesis: CKD alters the activity of individual CYPs responsible for vitamin D metabolism, leading to modified clearance of cholecalciferol.

ELIGIBILITY:
Inclusion criteria for CKD patients:

* vitamin D deficient (<30 ng/mL)
* hemoglobin >10 g/dL
* willing to abstain from fruit juices or alcohol within 7 days of PK assessments
* no changes in prescription or nonprescription medications within 4 wks of study start
* age 18-70 yrs
* If a diagnosis of CKD, must be due to diabetes mellitus or hypertension
* Signed informed consent

Inclusion Criteria for Healthy Controls:

* vitamin D deficient (<30 ng/mL)
* hemoglobin >10 g/dL
* willing to abstain from fruit juices or alcohol within 7 days of PK assessments
* no changes in prescription or nonprescription medications within 4 wks of study start
* age 18-70 yrs
* Signed informed consent

Exclusion criteria for CKD patients:

* History of >14 alcoholic drinks/wk
* Not likely to be compliant with study visits
* Pregnant or lactating
* Predisposition to or history of hypercalcemia
* History of allergy, sensitivity, or contraindication to probe drugs (seizures, drug metabolism interactions, etc)
* Use of prescribed or nonprescribed therapies that could interact with probe drugs (including prototypical inhibitors or inducers)
* Active autoimmune disease or active/recent infections requiring antimicrobial treatment within the previous 4 wks will be excluded to minimize inflammatory-mediated changes in vitamin D status and patient heterogeneity.
* Presence of clinically significant hepatic insufficiency (total bilirubin greater than 1.5 times the upper limit of normal or transaminase (ALT, AST) elevations greater than 2 times the upper limit of the laboratory reference range or liver disease
* Active seizure disorder or those patients receiving large doses of medications that are known to reduce seizure threshold
* Currently receiving cholecalciferol or a vitamin D analogue

Exclusion Criteria for Healthy Controls:

* History of >14 alcoholic drinks/wk
* Not likely to be compliant with study visits
* Pregnant or lactating
* Predisposition to or history of hypercalcemia
* History of allergy, sensitivity, or contraindication to probe drugs (seizures, drug metabolism interactions, etc)
* Use of prescribed or nonprescribed therapies that could interact with probe drugs (including prototypical inhibitors or inducers)
* Active autoimmune disease or active/recent infections requiring antimicrobial treatment within the previous 4 wks will be excluded to minimize inflammatory-mediated changes in vitamin D status and patient heterogeneity.
* Presence of clinically significant hepatic insufficiency (total bilirubin greater than 1.5 times the upper limit of normal or transaminase (ALT, AST) elevations greater than 2 times the upper limit of the laboratory reference range or liver disease
* Active seizure disorder or those patients receiving large doses of medications that are known to reduce seizure threshold
* Currently receiving cholecalciferol or a vitamin D analogue
* Any clinical evidence of chronic kidney disease as defined by the National Kidney Foundation Dialysis Outcomes Quality Initiative (NKF DOQI) guidelines

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-10; Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Change in area under the plasma concentration time curves for probe drugs (bupropion, midazolam, olmesartan and fexofenadine) from baseline to 12 weeks. | 12 weeks
  Change in area under the plasma concentration time curves for probe drugs (bupropion, midazolam, olmesartan, and fexofenadine) at 12 weeks.

SECONDARY OUTCOMES:
Change in area under the plasma concentration time curves for cholecalciferol from baseline to 12 weeks. | 12 weeks
  Change in area under the plasma concentration time curves for cholecalciferol at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Joy, PharmD, PhD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado, Aurora, Colorado
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No